CLINICAL TRIAL: NCT00527683
Title: Double-Blind, Randomized, Placebo- Controlled Trial of Vigabatrin for Short Term Abstinence From Cocaine in Cocaine Dependent Parolees
Brief Title: Double Blind Study of Vigabatrin for the Treatment of Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Catalyst Pharmaceuticals, Inc. (Industry)
Responsible Party: Jonathan D. Brodie, PhD, MD, Professor, Dept. of Psychiatry, New York University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H06-152
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Cocaine Dependence
Keywords: vigabatrin; GVG; addiction; treatment; cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive | interventions — Vigabatrin; Psychotherapy, Group

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Subjects will receive vigabatrin in escalating doses to 3 grams per day over three weeks, continued for 4 weeks and then tapered to zero over the next 2 weeks.
  Interventions: Drug: Vigabatrin; Behavioral: Group therapy
- B (Placebo Comparator): Orange juice and administration identical to Arm A.
  Interventions: Drug: Placebo; Behavioral: Group therapy

INTERVENTIONS:
Drug: Vigabatrin — crystalline drug dissolved in orange juice, dosage escalates from 500 mg twice daily to 1.5 g twice daily over a 3 week period. This dose is maintained for 4 weeks and then tapered to zero over the next two weeks
  Other Names: Sabril; CPP 109; gamma vinyl GABA; GVG
  Arms: A
Drug: Placebo — orange juice is administered twice daily in containers indistinguishable from the treatment arm.
  Arms: B
Behavioral: Group therapy — Participants attend group sessions once a week

SUMMARY:
The primary objective of this study is to assess the efficacy of vigabatrin for the treatment of cocaine dependence, based on the twice-weekly qualitative urine toxicologies for cocaine. Based on two prior unblinded human studies and 15 years of animal studies, this 100 subject double- blind, randomized study is designed to show if with vigabatrin treatment but not placebo, even non-hospitalized cocaine dependent individuals with ready access to cocaine will become cocaine abstinent if they are self motivated to stop their cocaine habit. To accomplish this, cocaine dependent subjects will be randomly assigned to either a placebo or vigabatrin treatment group and treated for a nine week period. The primary hypothesis is that as compared to the placebo arm, the vigabatrin treatment arm will show a significant increase in the number of subjects who are abstinent for the final 3 weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in the study, subjects must

* Be at least 18 years of age and no older than 55 years of age.
* Weigh more than 100 pounds.
* Have a DSM-IV diagnosis of cocaine dependence.
* Be seeking treatment for cocaine dependence.
* Have a urine sample positive for qualitative cocaine toxicology at initial screening.
* Have the ability to understand, and having understood, provide written informed consent to comply with the treatment protocol.
* Have a history and brief physical examination that demonstrate no clinically significant contraindication for participating in the study, in the judgment of the admitting physician and the Principal Investigator.
* Have normal, or, if necessary, corrected visual acuity, visual fields, and normal fundoscopy findings

Exclusion Criteria:

* In order to participate in the study, subjects must not:

  * Meet DSM-IV criteria for current dependence on any psychoactive substance other than cocaine, alcohol, nicotine, or marijuana or physiological dependence on alcohol requiring medical detoxification.
  * Have neurological or psychiatric disorders such as: psychosis, bipolar illness, major depression, organic brain disease, dementia, any disorder which would require ongoing treatment or which would make study agent compliance difficult, history of suicide attempts assessed and/or current suicidal ideation/plan.
  * Have serious medical illnesses or other potentially life threatening or progressive medical illness other than addiction that may compromise subject safety or study conduct.
  * Have a history of traumatic head injury.
  * Be mandated by a court to obtain treatment for cocaine dependence.
  * Have been treated for cocaine addiction, or abstained from cocaine use for a significant period, within the 6 months preceding screening.
  * Be unable to complete the study protocol because of probable incarceration or relocation from the clinical area.
  * Have AIDS (although AIDS is an exclusion criterion, a positive antibody titer to HIV is not).
  * Have active syphilis that has not been treated or refuse treatment for syphilis
  * Have a history of neuroleptic malignant syndrome.
  * Have known or suspected hypersensitivity to vigabatrin or any other GABAergic drug.
  * Have received a drug with known potential for toxicity to a major organ system within 30 days prior to study entry (e.g., isoniazid, methotrexate).
  * Have participated in any experimental study within 4 weeks, or participated in any clinical trial utilizing vigabatrin.
  * Be pregnant or lactating.
  * Have any clinically significant abnormal laboratory value.
  * Have had electroconvulsive therapy with the 3 months preceding screening.
  * Have had any opiate-substitutes (methadone, LAAM, buprenorphine) within 2 months preceding screening.
  * Have a history of i.v. cocaine (or other psychoactive drug) use within 2 months preceding screening.
  * Have a current or past history of seizure disorder, including alcohol- or stimulant related seizure, febrile seizure, or significant family history of idiopathic seizure disorder.
  * Have a visual field defect, or factor predisposing to visual field defects, including glaucoma, severe myopia, retinal disorder, cataracts, diabetes or uncontrolled hypertension.
  * Have my illness, condition, and use of medications, in the opinion of the Principal Investigator and the admitting physician, which would preclude safe or successful completion of the study.
  * Be using vigabatrin or any medication that could interact adversely with vigabatrin administration, based on the longest time interval of A or B below:

    * A) Five half-lives of other medication or active metabolite(s), whichever is longer;
    * B) Two weeks.
  * Be lactose intolerant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Three consecutive weeks of negative urine tests (benzoyl ecgonine) for cocaine use (no slips allowed). | These must be the last three weeks (7,8,9) of the trial.

SECONDARY OUTCOMES:
3 consecutive weeks of negative urines (one slip allowed) | Last 3 weeks (7,8,9) of the trial
cocaine craving | Weeks 1, 5,9

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Brodie, Ph.D., M.D., Principal Investigator — NYU Langone Health; Emilia Figueroa, M.D., Study Director — Clinica Integral de Tratamiento Contra las Adicciones, S.A de C.V.
Locations (1):
- Clinica Integral de Tratamiento Contra las Adicciones SA de CV, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Fechtner RD, Khouri AS, Figueroa E, Ramirez M, Federico M, Dewey SL, Brodie JD. Short-term treatment of cocaine and/or methamphetamine abuse with vigabatrin: ocular safety pilot results. Arch Ophthalmol. 2006 Sep;124(9):1257-62. doi: 10.1001/archopht.124.9.1257. PMID 16966620
- [Background] Brodie JD, Figueroa E, Laska EM, Dewey SL. Safety and efficacy of gamma-vinyl GABA (GVG) for the treatment of methamphetamine and/or cocaine addiction. Synapse. 2005 Feb;55(2):122-5. doi: 10.1002/syn.20097. PMID 15543630
- [Background] Brodie JD, Figueroa E, Dewey SL. Treating cocaine addiction: from preclinical to clinical trial experience with gamma-vinyl GABA. Synapse. 2003 Dec 1;50(3):261-5. doi: 10.1002/syn.10278. No abstract available. PMID 14515344
- [Derived] Brodie JD, Case BG, Figueroa E, Dewey SL, Robinson JA, Wanderling JA, Laska EM. Randomized, double-blind, placebo-controlled trial of vigabatrin for the treatment of cocaine dependence in Mexican parolees. Am J Psychiatry. 2009 Nov;166(11):1269-77. doi: 10.1176/appi.ajp.2009.08121811. Epub 2009 Aug 3. PMID 19651710